CLINICAL TRIAL: NCT04783597
Title: Early Prediction of Preeclampsia Using arteriaL Stiffness in High-risk prEgnancies; a Multinational Study (PULSE)
Brief Title: Early Prediction of Preeclampsia Using arteriaL Stiffness in High-risk prEgnancies
Acronym: PULSE
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Université de Montréal (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); University of British Columbia (Other); University of Glasgow (Other); Laval University (Other); Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government); McGill University (Other)
Responsible Party: Principal Investigator, Dr. Stella Daskalopoulou, Associate Professor - Department of Medicine, Division of Internal Medicine and Division of Experimental Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: MP-37-6854
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: High Risk Pregnancy; Arterial Stiffness; Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Vascular Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected from participants for serum and plasma biomarker analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Arterial Stiffness and Wave Reflection — Arterial stiffness and wave refection, a non-invasive test, will be collected and combined with standard clinical markers (blood biomarkers, ultrasound imaging) as well as medical and psychosocial questionnaires in order to test a comprehensive, multi-marker approach for pre-eclampsia prediction in high risk pregnant women.

SUMMARY:
Despite advances in obstetric care, preeclampsia (PE) remains the leading cause of maternal death and disability in both developed and developing countries, contributing to over 70,000 maternal and 500,000 fetal deaths annually worldwide. PULSE was designed using a preventative medicine approach, focusing on improving early detection of PE as opposed to managing symptoms after onset. The study aims to uncover the earliest possible signs of PE using a combination of novel clinical tools and established diagnostic techniques to better identify, track, and manage high risk pregnant women. Specifically, PULSE will be examining the incorporation of a non-invasive test for the measurement of arterial stiffness, which has been shown to be predictive of hypertensive disorders. This test, in combination with a wide range of blood biomarkers, detailed ultrasound imaging, and a comprehensive battery of physical and mental health questionnaires, represents the largest, most comprehensive preventative PE study to date. The results of this work has the potential to revolutionize the way PE and other hypertensive disorders of pregnancy are managed and treated and can serve to inform the design of future preventative clinical research studies.

DETAILED DESCRIPTION:
Existing predictive tools for preeclampsia (PE), including clinical characteristics, blood pressure, blood biomarkers, and uterine artery Doppler indices, have, at best, moderate predictive properties. While maternal symptoms often resolve with the delivery of the placenta, the burden of PE extends beyond pregnancy; afflicted women are at 3.1-fold increased odds of developing hypertension and 2.3-fold increased odds for cardiovascular disease later in life compared to women with uncomplicated pregnancies. Placental pathogenic changes associated with PE occur weeks to months before clinical manifestations develop, presenting a window of opportunity to identify early those women who will develop PE. The goal of the study investigators is to capitalize on this window and develop strategies for early prediction of PE.

As a composite measure of vascular health, measurement of arterial stiffness and wave reflection could represent a promising non-invasive tool for PE prediction. This multi-national 5-year observational prospective study aims to recruit 2400 participants across 8 sites in Canada, the US, and the UK. Participants will undergo 2 assessments, one in the first trimester (10 - 13 weeks gestation) and one in the second trimester (18 - 21 weeks gestation), which involve vascular measurements (arterial stiffness, blood pressure), blood sample collection, psychosocial and demographic questionnaires, and Uterine Artery Doppler imaging (only at second visit). Post-natal outcome measurements will be collected via medical charts for each participant 6-8 weeks post-partum. The primary objective of the study is to determine if, and to what extent, arterial stiffness and wave reflection parameters improve early prediction of PE beyond that achieved by currently available predictors in high-risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Presence of at least 1 high-risk factor or 2 moderate-risk factors for pre-eclampsia

Exclusion Criteria:

* >14 weeks gestation
* Multiple pregnancy
* History of heart disease, stroke, or peripheral arterial disease
* Infectious diseases/conditions, such as Hepatitis B/C, HIV, and COVID19

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women at high risk of developing preeclampsia
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of pre-eclampsia | up to 6 weeks post-partum (after delivery)
  According to the Society of Obstetricians and Gynaecologists (SOGC) guidelines, upon the presence of 2 criteria: 1) hypertension; chronic (pre-dating pregnancy or diagnosed <20 weeks' gestation) or de novo/gestational (diagnosed ≥20 weeks') hypertension along with 2) de novo end-organ dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Stella S Daskalopoulou, MD, PhD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No